CLINICAL TRIAL: NCT01805986
Title: Investigation of Grey Matter Pathology Using Ultra High Field (7T) MRI Scanner
Brief Title: Investigation of GM Pathology Using Ultra High Field (7T) MRI Scanner
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 12115; 13920 (Other: Clinical Research Network); 12/EM/0452 (Other: NRES); 917 (Other Grant/Funding Number: MS Society)
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, other neurological conditions
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MS patient

SUMMARY:
Magnetization transfer imaging is a magnetic resonance technique that has been used over the last few years, and known for its ability to detect abnormalities that can be difficult to detect by conventional MRI techniques.

The investigators would like to test if using an 7 Tesla MRI research scanner can help us diagnose Multiple Sclerosis more efficiently compared to the current clinical practice, i.e. if Multiple Sclerosis lesions in Gray Matter can be more readily identified and associated with disease stage on Magnetic Transfer MRI images as opposed to conventional procedures. Image analysis will allow the investigators to perform lesion segmentation and sequence comparison between different MRI techniques. The investigators will apply computation techniques to measure the local cortical thickness. Repeated scans at 6 monthly intervals over two years will give an insight into the changes in cortical thickness over time. Based on obtained data the investigators will look for the relationship between lesion loads in White Matter and Gray Matter, cortical thickness and disease stage.

DETAILED DESCRIPTION:
Purpose for this study:

This research group has previously investigated the usefulness of a powerful new MRI scanner and have found that the 7 Tesla MRI is able to provide detailed structural images of the cortex of the brain which can uncover pathology such as cortical demyelinating lesions in MS patients. Multiple sclerosis (MS) affects the grey matter as well as the white matter of the brain and spinal cord. However as white matter lesions are more easily visible both pathologically and on MRI, therefore most MS research has focused on white matter demyelination. The investigators would like to assess whether MS lesions in Gray Matter as well as White Matter can be more readily identified on Magnetic Transfer Ratio (MTR) images as opposed to standard protocols such as DIR, T2* and T1-weighted MPRAGE by comparing the results of the manual detection.

The investigators will correlate lesion loads against cortical thickness and both lesion loads and cortical thickness against disease state both globally and on a regional basis. The investigators will then compare averaged, normalized profiles from different cortical ribbon regions between patients and controls to determine whether a particular layer of the cortical strip is more affected. The investigators will also correlate Gray Matter changes with distant and neighboring White Matter lesions. In addition, the investigators will also build an average lesion map across all subjects, which can be compared against the results published in literature. The investigators will use the manual lesion maps to characterize the regions of the cortex that deviate from normally appearing Gray Matter.

How this project will be carried out:

The investigators will study patients with MS and other neurological disease, and patients who are followed already at the neurology. All patients would have had already a brain scan.

For comparison purposes the investigators will study healthy volunteers, in order to demonstrate that any new findings demonstrable with the 7T MRI scan are indeed related to pathology.

Ethical issues:

Occasionally the investigators discover incidental abnormalities on brain scans of those who participate in the study. In such circumstances the investigators will adhere to University of Nottingham Incidental Findings Procedure. In the Participant Information Sheet the investigators will explain that if the investigators notice any abnormality on MR scans (for healthy volunteer) or abnormality on MR scan not expected to be seen under patient's neurological diagnosis (for patients) the investigators will refer them to their GP. The investigators will send a letter to patient's GP informing that the investigators have detected a possible abnormality on the scan. The investigators will show the scans to a radiologist based in Academic Radiology at the QMC, who will contact participant's GP if further action is required.

ELIGIBILITY:
Inclusion criteria:

* Patients with MS or other neurological disease which already had at least 1 MRI scan.
* Healthy volunteers which had no indication of neurological disease in the past.
* Do not have significant cognitive impairment and are able to give consent.
* Will not have any contraindication for MR imaging

  * Are able to lie flat for up to 60 mins.
  * Age 25 and over.

Exclusion criteria:

* Pregnancy
* Have any implants in the body.
* Have aneurysm clips.
* Have pacemaker or artificial heart valve.
* Have foreign bodies in their body (e.g. shrapnel).

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients studied will be those with known MS. For purposes of comparison as described previously, we will also seek to include healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
The number of Gray Matter lesions detected using different sequences. | 2 years

SECONDARY OUTCOMES:
Comparison of MRI sequencies | 2 years
  To determine whether Magnetisation Transfer Ratio (MTR) maps are more sensitive for detection of cortical lesions than Double Inversion Recovery (DIR), T2* and phase maps, or Magnetisation Prepared Rapid Acquisition Gradient Echo (MPRAGE) and to better characterise cortical lesions using a combination of sequences.
To determine the relationship between cortical thickness as measured on T1 weighted images and GM and WM lesion load. | 2 years
Regional variation in the brain | 2 years
  To determine the origins of regional changes previously detected via voxel based analysis and histogram analysis, using a multiscale approach, working down from identifying regional variations across the cortex, to identifying whether regional changes are associated with changes in so called Normal Appearing White Matter (NAGM), or whether they are associated with diffuse or focal GM lesions.
To detect cortical variations in MT inside and outside GM lesions, in a longitudinal pilot study, reflecting possible cortical remyelination. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, PhD, Principal Investigator — University of Nottingham